CLINICAL TRIAL: NCT06082271
Title: Comparative, Randomized Study on the Anti-inflammatory and Regenerative Efficacy of a New Medical Device (DM) Based on Hydrolyzed Collagen Peptides in Patients With Femoro-acetabular Impingement Undergoing Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Eleonora Olivotto (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAI_DM
Record Dates: First submitted 2023-09-21; First posted 2023-10-13 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Femoroacetabular Impingement; Hip Arthroscopy; Hip Osteoarthritis; Hydrolyzed Collagen Peptides
MeSH Terms: conditions — Femoracetabular Impingement; Osteoarthritis, Hip | interventions — Cortisone

STUDY DESIGN:
Intervention Model Description: Patients scheduled for hip arthroscopy for treatment of FAI and/or labral pathology were enrolled. The two treatments, cortisone (gold standard) or collagen Pepetids, were administrated to patients intraoperatively with random sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cortisone (C) (Active Comparator): To improve the outcome of the arthroscopy during the procedure, cortisone is injected for anti-inflammatory purposes at the end of the surgical procedure.
  Interventions: Drug: Cortisone
- Hydrolyzed Collagen Peptides (Experimental): The use is alternative to cortisone
  Interventions: Device: Class III medical Hydrolyzed Collagen Peptides PEP-52 (Peptys)

INTERVENTIONS:
Device: Class III medical Hydrolyzed Collagen Peptides PEP-52 (Peptys) — Anti-inflammatory and regenerative effect, 5 mg/ml
  Arms: Hydrolyzed Collagen Peptides
Drug: Cortisone — DEPO-MEDROL 40 mg/ml + 1 cc di NAROPINA 0,75% 7,5 mg/ml
  Arms: Cortisone (C)

SUMMARY:
Hip Osteoarthritis (HOA) is the most common joint disorder and a major cause of disability in the adult population. Thus, the early diagnosis, prevention, and treatment of the early stages of the disease and of the pre-arthritic condition, in particular in adolescents and young adults, is crucial to reducing the incidence of end-stage HOA and the need for total hip replacement (THR).

Evidence has mounted for a prominent etiologic role of femoroacetabular impingement (FAI) in the development of early HOA leading to the development of early cartilage and labral damage in the non-dysplastic hip. Therefore, the surgical treatment of FAI with mini-invasive arthroscopy is crucial. To improve the outcome after surgery, cortisone is routinely injected during the procedure for anti-inflammatory purposes.

The aim of the study is to compare the use of cortisone (gold-standard) (C) to a new class III medical device based on hydrolysed Collagen Peptides PEP-52, Peptys (P) and to investigate potential associations among the preoperative symptoms and hip function, the outcomes after arthroscopic surgery and biomarkers in synovial fluids (SFs).

DETAILED DESCRIPTION:
Patients scheduled for hip arthroscopy for treatment of FAI and/or labral pathology will be enrolled. The two treatments, C or P, will be administrated to patients with random sampling. SFs samples, when available, are obtained by aspiration just prior to surgical intervention, collected and stored for biomarkers analysis.

At the baseline, OA severity will be assessed with a radiographic scoring system (Tönnis classification). Physical examination and clinical assessment using the Hip disability & Osteoarthritis Outcome Score (HOOS) and VAS score for pain will be performed at the time of surgery and at 1-6 months of follow up. At the time of surgery, chondral (Outerbridge score) and labral pathology based on direct arthroscopic visualization will be also evaluated.

The presence of inflammatory molecules at the baseline in the SFs will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* candidates for hip arthroscopy for femoroacetabular impingement (FAI)
* ability to provide informed consent

Exclusion Criteria:

* inability to provide informed consent;
* patients suffering from cancer or with poor general health conditions;
* patients suffering from coagulation diseases;
* positive history of tumor, infection, rheumatic or metabolic disease in the joint undergoing surgery;
* systemic inflammatory rheumatic diseases;
* pregnant or breastfeeding women;
* patients with proven hypersensitivity to collagen of bovine origin or vitamin C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Hip disability & Osteoarthritis Outcome Score (HOOS) has five domains (pain, symptoms, activities of daily living, sports, recreational activities, quality of life): higher scores better hip function. | Pre-operative; 1 and 6 months post-operative
  Investigate the preoperative symptoms and hip function
Visual Analogue Scale (VAS) | Pre-operative; 1 and 6 months post-operative
  Investigate the preoperative hip pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain.
Osteoarthtitis severity assessed with radiographic scoring system (Tönnis classification) | Pre-operative; 1 and 6 months post-operative
  Investigate the degenerative changes to the hip. The score consists of three progressive degrees: 0 no osteoarthritis; form 1 to 3 increasing the degeneration.

SECONDARY OUTCOMES:
Correlation between biomarkers in the pre-operative synovial fluid/urine and post-operative outcomes | Pre-operative; 1 and 6 months post-operative
  Evaluation of the correlation between the presence of inflammatory molecules in the pre-operative synovial fluid and the post-operative HOOS in both groups and the presence of collagen degradation products in the urine in the pre-operative
Correlation between biomarkers in the pre-operative synovial fluid/urine and post-operative pain | Pre-operative; 1 and 6 months post-operative
  Evaluation of the correlation between the presence of inflammatory molecules in the pre-operative synovial fluid and the post-operative pain score VAS in both groups and the presence of collagen degradation products in the urine in the pre-operative
Differences between the two study groups | 6 months post-operative
  Evaluate the differences between group I and group I+P in the clinical and functional outcome and in the use of analgesics

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nepple JJ, Clohisy JC; ANCHOR Study Group Members. Evolution of Femoroacetabular Impingement Treatment: The ANCHOR Experience. Am J Orthop (Belle Mead NJ). 2017 Jan/Feb;46(1):28-34. PMID 28235110
- [Background] Agricola R, Heijboer MP, Bierma-Zeinstra SM, Verhaar JA, Weinans H, Waarsing JH. Cam impingement causes osteoarthritis of the hip: a nationwide prospective cohort study (CHECK). Ann Rheum Dis. 2013 Jun;72(6):918-23. doi: 10.1136/annrheumdis-2012-201643. Epub 2012 Jun 23. PMID 22730371
- [Background] Goldring MB, Otero M. Inflammation in osteoarthritis. Curr Opin Rheumatol. 2011 Sep;23(5):471-8. doi: 10.1097/BOR.0b013e328349c2b1. PMID 21788902
- [Background] Sellam J, Berenbaum F. The role of synovitis in pathophysiology and clinical symptoms of osteoarthritis. Nat Rev Rheumatol. 2010 Nov;6(11):625-35. doi: 10.1038/nrrheum.2010.159. Epub 2010 Oct 5. PMID 20924410
- [Background] Scanzello CR, Goldring SR. The role of synovitis in osteoarthritis pathogenesis. Bone. 2012 Aug;51(2):249-57. doi: 10.1016/j.bone.2012.02.012. Epub 2012 Feb 22. PMID 22387238
- [Background] Berenbaum F. Osteoarthritis as an inflammatory disease (osteoarthritis is not osteoarthrosis!). Osteoarthritis Cartilage. 2013 Jan;21(1):16-21. doi: 10.1016/j.joca.2012.11.012. Epub 2012 Nov 27. PMID 23194896
- [Background] Nepple JJ, Carlisle JC, Nunley RM, Clohisy JC. Clinical and radiographic predictors of intra-articular hip disease in arthroscopy. Am J Sports Med. 2011 Feb;39(2):296-303. doi: 10.1177/0363546510384787. Epub 2010 Nov 23. PMID 21098820
- [Background] Patel K, Wallace R, Busconi BD. Radiology. Clin Sports Med. 2011 Apr;30(2):239-83. doi: 10.1016/j.csm.2010.12.004. PMID 21419955
- [Background] Dolan MM, Heyworth BE, Bedi A, Duke G, Kelly BT. CT reveals a high incidence of osseous abnormalities in hips with labral tears. Clin Orthop Relat Res. 2011 Mar;469(3):831-8. doi: 10.1007/s11999-010-1539-6. Epub 2010 Oct 1. PMID 20886325
- [Background] Simpson J, Sadri H, Villar R. Hip arthroscopy technique and complications. Orthop Traumatol Surg Res. 2010 Dec;96(8 Suppl):S68-76. doi: 10.1016/j.otsr.2010.09.010. Epub 2010 Oct 30. PMID 21036688
- [Background] Volpi P, Zini R, Erschbaumer F, Beggio M, Busilacchi A, Carimati G. Effectiveness of a novel hydrolyzed collagen formulation in treating patients with symptomatic knee osteoarthritis: a multicentric retrospective clinical study. Int Orthop. 2021 Feb;45(2):375-380. doi: 10.1007/s00264-020-04616-8. Epub 2020 May 23. PMID 32447428
- [Background] Krych AJ, Griffith TB, Hudgens JL, Kuzma SA, Sierra RJ, Levy BA. Limited therapeutic benefits of intra-articular cortisone injection for patients with femoro-acetabular impingement and labral tear. Knee Surg Sports Traumatol Arthrosc. 2014 Apr;22(4):750-5. doi: 10.1007/s00167-014-2862-3. Epub 2014 Feb 1. PMID 24488223